CLINICAL TRIAL: NCT04242888
Title: The Acute Effects of Pragmatic Manual Therapy on the Range of Motion of Shoulder Joint
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Isra University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 1602-PhD-001
Record Dates: First submitted 2020-01-14; First posted 2020-01-27 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Shoulder Impingement; Prehabilitation; Rehabilitation
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Intervention Model Description: Four trial of a single group quasi experimental design on healthy subjects through individual intervention followed by similar trial on subject with shoulder pathology through combination of all intervention.
Who Masked: Participant, Outcomes Assessor
Masking Description: participant and outcome assessor does not know the purpose of the trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Rotator Cuff Facilitation (Experimental): The function of Rotator cuff muscles is passively augmented in one of the 5 trials
  Interventions: Other: pragmatic manual therapies
- Serratus Anterior Stretch (Experimental): Seratus anterior muscles is stretched through a novel technique
  Interventions: Other: pragmatic manual therapies
- Posterior Capsular Stertch (Experimental): Posterior capsule is stretched through a novel maneuver
  Interventions: Other: pragmatic manual therapies
- Acromioclavicular Joint Mobilization (Experimental): Acromio clavicular joint is mobilized posterio-anterior
  Interventions: Other: pragmatic manual therapies
- Pragmatic Interventions (Experimental): The pragmatic interventions is a set of interventions which include
  1. Rotator cuff facilitation
  2. Posterior capsular stretch
  3. Serratus anterior muscle stretch
  4. Acromioclaicualr joint mobilization
  5. Thoracic spine manipulation and
  6. Stretch to the subclavious muscles
  Interventions: Other: pragmatic manual therapies

INTERVENTIONS:
Other: pragmatic manual therapies — three of the intervention are novel and the rest of the interventions are in practice but seldom used to treat the shoulder disorder.
  Other Names: Rotator cuff facilitation; Serratus anterior stretch; Acromioclavicular joint mobilization; Posterior capsular stretch; A set of pragmatic interventions

SUMMARY:
Current studies on the mechanism of subacromial impingement and other shoulder pathology reveal that multiple factors are responsible for impingement. These include serratus anterior dysfunction, rotator cuff insufficiency, posterior capsular tightness, acromioclavicular joint, thoracic spine stiffness and extensibility of the pectoralis minor and subclavius muscles. Manual intervention should therefore address these issues in conjunction with the other therapies. Novel interventions have been designed pilot tested for each of these factors to produce a healing environment. The purpose of this study is to evaluate the effects of each individual factor and combination of all on the range of motion of shoulder joint in healthy subjects and subjects with a restricted range of motion of shoulder joint respectively. The subject will be allocated randomly into four groups with respect to objective 1 and each of the groups will be evaluated as a quasi-experiment design (pretest-posttest) for healthy each of 30 subjects. Beneficial intervention among the four trials and other previously reported beneficial in improving the shoulder joint range will be combined in and termed as pragmatic intervention protocols. Pragmatic interventions on subjects with the restricted range in shoulder pathology will be tested through a similar design. The effects of these interventions on the Quality of life measured through the Urdu version of Shoulder pain and disability in subjects with shoulder pathology will also be tested.

DETAILED DESCRIPTION:
Shoulder disorders are the 3rd commonest among musculoskeletal conditions. Its prevalence is estimated 7-26% at one point of time and 67% of the individuals experience shoulder pain once in their life. Subacromial impingements (SAIS) are the frequent diagnosis accounting for 45-65% of all shoulder disorders. It is defined as "a condition in which the tendons of the rotator cuff muscles, long head of the biceps or the subacromial bursa are entrapped between the humeral head inferiorly and anterior acromion superiorly.

Multiple researchers have studied interventions which affect the shoulder range of motions. Thoracic spine manipulation improves the shoulder range of motion. Similarly, Stretching the pectorallis minor muscles improve shoulder kinematics. Manual intervention for subscapularis, infra spinatus, and serratus anterior are non-existent to investigators' knowledge. Modification to stretch the posterior capsule in a pragmatic manner is described and recommended but trials are nonexistent. Acromioclavicular joint being the part of the scapolo-glenohumeral complex has a role to play in the kinematics of the shoulder but trials on its mobilization with respect to shoulder range of motion are not been studies. These gaps in research in relation to understanding of the mechanism of shoulder pathology and subsequent intervention are also identified but trials and interventions are non-existent.

The understanding of the complex relations of the intrinsic and extrinsic factors necessitates the development of manual therapy interventions to address the factors which are adversely affect range of motion of shoulder joint. The purpose of this research is to develop and propose manual therapy interventions for shoulder joint which can effectively address the limitations in shoulder joint ranges of motion in both healthy subjects and subjects with shoulder pathology having decrease range of motion through a series of primitive trials.

AIMES AND OBJECTIVES The primary purpose of this study is to evaluate the short term effects of Pragmatic manual interventions on range of motion of the shoulder joint in healthy individual and individuals with shoulder pathology who have restricted ranges of motion .The aims of this study are therefore to

1. To evaluate the effects of pragmatic interventions in healthy asymptomatic subjects with respect to the changes in shoulder joint restricted range of motion
2. To evaluate the effects of interventions in symptomatic shoulder individual with restriction in their shoulder range of motion and short term change in the shoulder related quality of life and pain MATERIAL AND METHOD A single group quasi-experimental (pretest-posttest) design will be used for all the trials in this study. It will be conducted at Helping Hand Institute of Rehabilitation Sciences, Mansehra. The study will be composed of 4 trials in the first phase on healthy subject with respect to each of the proposed pragmatic (novice) intervention consistent with the first objective and exploratory in nature. Subjects will be randomly allocated to the initial four groups. The initial 4 trials on healthy subjects are chosen since the effects of each of the proposed pragmatic interventions is not been studied but advocated. Healthy subjects with restriction in shoulder ROM are deemed appropriate since other confounding factors such as pain is absent and objectives could be achieved. In Phase 2, trial on patient with shoulder pathology will be conducted after evaluating the effects on range of motion in healthy individual. Each trial will recruit 30 subjects. subjects in trial 5 with shoulder pathology will be assessed through Urdu version of shoulder pain and disability index at baseline, after one week and 5 weeks of pragmatic interventions. A sample size of 30 for each trial ( a total of 150 subject) is deemed appropriate after a pilot trial on 5 healthy subject which produced a meaningful difference of 15 degree change in abduction, and 3 cm difference in reaching up behind the back and using standard deviation estimates from previous studies. Finally, The urdu translated and validated version of SPADI will used to measure shoulder related pain and Disability. Ethical approval will be sought from REC Isra university and Ethical committee of HHIRS. Subjects consent will be taken in writing (annex 2) and full study information will be given (annex 3). Each of Phase 1 and phase 2 of this study will be completed in 6 months (a total of 1 year) from August 2019 to August 2020.

SUBJECTS ASSESSMENT PROCEDURE For healthy subject of the initial 4 trials, subjects willing to participate will be screened against the inclusion and exclusion criteria. Each participant for trial 5 with shoulder pathologies will be assessed thoroughly and screened against the inclusion and exclusion criteria. Demographic information, information related to history of the presenting complaint, past medical and surgical history, hobbies, occupation, drug history and social history will be collected from all the eligible subjects in trial 5. Additional information in relation to date of onset, behavior of symptoms, aggravating, easing factors, previous treatment including injection and other surgical interventions, relevant investigation will be collected.

A detailed objective examination process will be followed for participants in trial 5. Examination process will include inspection of the shoulders, cervical spine and thoracic spine from the front, each side and back. Any abnormality seen will be documented.

Inspection will be followed by ruling out any pathology of the neck by asking the patient to perform active neck rotation to each side, side flexion, extension and flexion and any pain, discomfort and paraesthesia will be noted. These quick movements are assumed sufficient to rule out any pathology of the neck. Neck movements will be followed by the active elevation (flexion and abduction) of the shoulder joint and any pain, restriction in range and willingness to movement will be noted. Active reaching behind the back will be performed and any limitation in comparison with the asymptomatic side noted. Limitation will be measures from the respective posterior superior iliac spine though measuring tape. Active elation of the arm is followed by the passive movements of abduction, flexion, and medial rotation. Any limitation of range, end feel and pain will be noted during each of the passive movement. Active resisted movement of abduction, medial rotation, later rotation of shoulder and flexion and extension of elbow are followed and strength/pain will be noted. The systematic procedure of assessment followed from Cyriax and has been found highly reliable(39) and assessment procedure including similar procedures Special test such as Neer's sign, Hawkin kennedy test, scarf test, speed test, O'brien's test will be administered to determine SAIS.

ELIGIBILITY:
Inclusion Criteria:

* For trial 1-4

  1. Limitation in Abduction or Internal rotation or reaching behind up or down the back
  2. A score of 1 and 2 on FMS For trial 5
* main complaint in gleno-humeral joint
* Limitation in Range of motion of Abduction or internal rotation or external rotation or reaching up behind the back or reaching down behind down the neck , all or only one of the limitation in comparison with the unaffected joint.

Exclusion Criteria:

* For trial 1-4

  1. Any known pathology or deformity of the shoulder joint
  2. A zero and 3 score on FMS For trial 5

  <!-- -->

  1. Previous history of dislocation or fracture in shoulder
  2. Severe underlying chronic medical condition
  3. shoulder surgeries
  4. Brachial plexus and axillary nerve injuries
  5. Severe constant shoulder pain which does not fit into the inclusion criteria
  6. Pain associated with shoulder swelling, redness or cysts
  7. Known rheumatoid arthritis
  8. Steroid injection within two weeks
  9. Psychosocial yellow flags or intellectual disability

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-09-02 (Actual); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Shoulder External Rotation | 12 months
  The change in external rotation range will be assessed at baseline and soon after the application of intervention in each of the trial. A higher score indicate improvement. A digital inclinometer will be used for measurement.
Shoulder Internal Rotation | 12 months
  The change in internal rotation range will be assessed at baseline and soon after the application of in each of the trial.A higher score indicate improvement. A digital inclinometer will be used for measurement.
Shoulder Abduction Range | 12 months
  The change in abduction range will be assessed at baseline and soon after the application of intervention in each of the trial.A higher score indicate improvement. A digital inclinometer will be used for measurement.
Shoulder Flexion | 12 months
  The change in Flexion range will be assessed at baseline and soon after the application of intervention in each trial. A higher score indicate improvement. A digital inclinometer will be used for measurement.
Reaching Up Behind the Back | 12 months
  The change in the distance between tip of the middle finger of one hand and the thumb of the other hand will be measured through measuring tap in each trial, as measured in functional movement screen.A lower difference between the scors indicates improvement.
Reaching Down Behind the Neck | 12 months
  the change in the distance between tip of the middle finger of one hand and the thumb of the other hand will be measured through measuring tap in each trial, as measured in functional movement screen.A lower difference between the scors indicates improvement.
Shoulder pain and Disability Index Urdu version | 12 months
  Change in scores Shoulder pain and disability index Urdu version will be assessed at baseline line in subjects with shoulder pathology and at 6th week of the combined intervention protocol. Less score indicate improved pain and disability

SECONDARY OUTCOMES:
Subject feed back questions | 12 months
  Suject feedback through a self construct subjective questionaire regarding various aspect of the intervention/interventions will be evaluate

CONTACTS AND LOCATIONS:
Locations (1):
- HHIRS, Mansehra, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No
Data will be available in two phases. work on the first part in progress and will be shared when available

REFERENCES:
- [Background] Seitz AL, McClure PW, Finucane S, Boardman ND 3rd, Michener LA. Mechanisms of rotator cuff tendinopathy: intrinsic, extrinsic, or both? Clin Biomech (Bristol). 2011 Jan;26(1):1-12. doi: 10.1016/j.clinbiomech.2010.08.001. Epub 2010 Sep 16. PMID 20846766
- [Background] Cools AM, Declercq G, Cagnie B, Cambier D, Witvrouw E. Internal impingement in the tennis player: rehabilitation guidelines. Br J Sports Med. 2008 Mar;42(3):165-71. doi: 10.1136/bjsm.2007.036830. Epub 2007 Dec 10. PMID 18070811
- [Background] Phadke V, Camargo P, Ludewig P. Scapular and rotator cuff muscle activity during arm elevation: A review of normal function and alterations with shoulder impingement. Rev Bras Fisioter. 2009 Feb 1;13(1):1-9. doi: 10.1590/S1413-35552009005000012. PMID 20411160
- [Background] Teyhen DS, Miller JM, Middag TR, Kane EJ. Rotator cuff fatigue and glenohumeral kinematics in participants without shoulder dysfunction. J Athl Train. 2008 Jul-Aug;43(4):352-8. doi: 10.4085/1062-6050-43.4.352. PMID 18668167
- [Background] Wilk KE, Hooks TR, Macrina LC. The modified sleeper stretch and modified cross-body stretch to increase shoulder internal rotation range of motion in the overhead throwing athlete. J Orthop Sports Phys Ther. 2013 Dec;43(12):891-4. doi: 10.2519/jospt.2013.4990. Epub 2013 Oct 30. PMID 24175603
- [Background] Chopp JN, O'Neill JM, Hurley K, Dickerson CR. Superior humeral head migration occurs after a protocol designed to fatigue the rotator cuff: a radiographic analysis. J Shoulder Elbow Surg. 2010 Dec;19(8):1137-44. doi: 10.1016/j.jse.2010.03.017. Epub 2010 Jul 3. PMID 20598916
- [Background] Kibler WB, Sciascia A. Current concepts: scapular dyskinesis. Br J Sports Med. 2010 Apr;44(5):300-5. doi: 10.1136/bjsm.2009.058834. Epub 2009 Dec 8. PMID 19996329
- [Background] Ekstrom RA, Donatelli RA, Soderberg GL. Surface electromyographic analysis of exercises for the trapezius and serratus anterior muscles. J Orthop Sports Phys Ther. 2003 May;33(5):247-58. doi: 10.2519/jospt.2003.33.5.247. PMID 12774999
- [Result] Keramat Ullah Keramat. Conservative treatment preferences and the plausible mechanism of Neer's stage 1 of shoulder impingement in younger people. J Pak Med Assoc. 2015 May;65(5):542-7. PMID 26028390
- [Result] Keramat KU, Mc Creesh K, Kropmans T. Voluntary Co-Contraction Exercise Effective In Early Stage Of Subacromial Impingement Syndrome Management. International Journal of Rehabilitation Sciences (IJRS). 2017;4(02):7-13.
- [Derived] Keramat KU, Naveed Babur M. Pragmatic posterior capsular stretch and its effects on shoulder joint range of motion. BMJ Open Sport Exerc Med. 2020 Sep 9;6(1):e000805. doi: 10.1136/bmjsem-2020-000805. eCollection 2020. PMID 33062302